## **DRCR Retina Network**

# Randomized Trial of Intravitreous Aflibercept Versus Intravitreous Bevacizumab + Deferred Aflibercept for Treatment of Center-Involved Diabetic Macular Edema (Protocol AC)

# **Statistical Analysis Plan**

| VERSION<br>NUMBER | AUTHOR | APPROVER | EFFECTIVE<br>DATE | REVISION DESCRIPTION |
|---|---|---|---|---|
| 1.0 | Wesley Beaulieu | Michele Melia | 02 Feb 2019 | Initial version for Protocol version 2.0 |
| 1.1 | Wesley Beaulieu | Michele Melia | 24 Apr 2020 | Increased upper limit of 2-year visit window due to COVID-19 pandemic. Implemented strategies for controlling the Type I error rate. Modified diabetic retinopathy progression scale per specifications from fundus photograph reading center. Made clarifications. Revisions were made prior to initial data analysis. Applies to Protocol version 3.0 |
| 1.2 | Wesley Beaulieu<br>Danni Liu | Maureen Maguire | 28 July 2021 | Added methods to control for multiplicity. Other minor changes. Revisions were made prior to initial data analysis. Applies to Protocol version 4.0. |
| 1.2 | Danni Liu | Maureen Maguire | 24 March 2022 | Minor changes and clarifications to Sections 3.3 and 4.0. |

| SIGNATURES |
|----------------------|
| AUTHOR |
| APPROVER |
| PROTOCOL<br>DIRECTOR |

### 1.0 Introduction

1

17

- 2 This document outlines the statistical analysis plan for the DRCR Retina Network protocol
- 3 comparing the anti-vascular endothelial growth factor (anti-VEGF) drug aflibercept versus
- 4 bevacizumab + deferred aflibercept for the treatment of center-involved diabetic macular edema
- 5 (CI-DME) in eyes with at least moderate vision loss (Protocol AC). Moderate vision loss is
- 6 defined as an Electronic-Early Treatment Diabetic Retinopathy Study (E-ETDRS) letter score of
- 7 68 to 24, which corresponds to an approximate Snellen equivalent of 20/50 to 20/320.
- 8 The primary objective of the protocol is to determine whether there is a treatment group
- 9 difference in mean change in visual acuity from baseline over two years (area under the curve
- 10 [AUC]). Participants will have visits every 4 weeks in year 1 and every 4 to 16 weeks in year 2,
- depending on the clinical course.
- 12 Study eyes will be assigned randomly to the two treatment groups in a 1:1 ratio. Participants may
- have one or two study eyes. Randomization of participants with one study eye will be stratified
- by site. Participants with two study eyes will have one eye randomized to each treatment,
- stratified by visual acuity of the eye with better visual acuity. If visual acuity is the same in both
- eyes, then the right eye will be considered to have better visual acuity than the left eye.

### 2.0 Primary Outcome Analysis

- 18 The primary analysis will consist of a treatment group comparison of mean change in visual
- acuity from baseline over two years adjusting for baseline visual acuity and the number of study
- eyes for the participant (one or two). Correlation arising from participants contributing two eyes
- 21 to the analysis will be modeled by including a random intercept term for participant using a
- 22 linear mixed effects model with robust variance estimation. The mathematical form of this model
- for eye i from participant j is as follows:

24 
$$AUC_{ij} = \beta_0 + \beta_1 \times BaselineVision_{ij} + \beta_2 \times NumEyes_j + \beta_3 \times Treatment_{ij} + u_i + \epsilon_{ij}$$

$$u_j \sim N(0, \sigma_{participant}^2)$$

26 
$$\epsilon_{ij} \sim N(0, \sigma^2)$$

- 27 The primary analysis is an intention-to-treat analysis. It will include all randomized eyes
- according to treatment group assignment at baseline. For each eye, AUC will be calculated by
- 29 the trapezoidal rule using the following formula:

30 
$$AUC = \sum_{i=1}^{n} \left( \frac{V_i + V_{i+1}}{2} \times (d_{i+1} - d_i) \right)$$

- Where  $V_i$  is the visual acuity measured at the  $i^{th}$  visit,  $d_i$  is the number of days from
- randomization to the  $i^{th}$  visit, and n is the number of outcome visits included in the analysis. For
- presentation, AUC will be divided by the number of days between baseline and the  $n^{th}$  visit so

- that the value shown will have units of letters rather than letter days (e.g., 728 days for the
- primary outcome at 104 weeks). This statistic can then be interpreted as the average change in
- visual acuity over the time between baseline and the  $n^{th}$  visit. All analysis visits will be included
- 37 for calculation of AUC and the number of days will be calculated based on the target date for the
- 38 visit: 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 68, 84, and 104 weeks (see Section 8.2 for a
- 39 description of analysis windows).
- 40 The P value, adjusted difference, and associated 95% confidence interval will be reported for the
- 41 treatment group effect. If the P value for the test of the treatment effect is less than or equal to
- 42 .05, then it will be concluded that there is a significant difference for change in visual acuity over
- 43 two years between the groups. In other words, if  $P \le .05$ , then the null hypothesis of  $\beta_3 = 0$  will
- 44 be rejected.

62

- 45 Markov Chain Monte Carlo (MCMC) multiple imputation with 100 imputations will be used to
- 46 impute missing data. The imputation will be performed separately for each treatment group and
- 47 the imputation model will include baseline visual acuity, change in visual acuity from baseline at
- all analysis visits, and the number of study eyes for the participant. Any imputed value outside of
- 49 the range for electronic visual acuity measurements (<0 or >100 letters) will be truncated at the
- closest measurable value (i.e., 0 or 100).
- A plot showing the change in visual acuity from baseline by treatment group over time will be
- 52 constructed using observed data. In general, summary statistics (e.g., within-group means and
- standard deviations), will be based on observed data while estimates from statistical models (e.g.,
- 54 treatment group differences, confidence intervals, and P values) will be based on imputed data.

### 2.1 Sensitivity Analyses

### 56 Complete Case Analysis

- A sensitivity analysis including only observed data from participants completing the 104-week
- visit (no imputation) will be conducted. If the analyses of imputed and observed data differ
- substantially, then exploratory analyses will be performed to evaluate factors that may have
- 60 contributed to the difference. The sensitivity analysis of completers will only be performed if
- more than 10% of randomized participants do not complete the 104-week visit.

### Tipping Point Analysis

- Multiple imputation assumes that data are missing at random (MAR). In the present study, this
- would mean that whether change in visual acuity is missing or observed may be a function of
- observed baseline characteristics included in the imputation model, but not a function of the
- unobserved follow-up data being imputed. This assumption cannot be tested directly since these
- data are unknown. However, a tipping point analysis will be conducted to adjust the imputed
- values using a shift parameter and thereby determine how severe the departure from MAR must
- be to change the outcome of the analysis with respect to rejecting or failing to reject the null
- 70 hypothesis.

- A shift parameter will be applied to the imputed values in the aflibercept group to determine the
- 72 tipping point at which the results of the primary analysis are nullified. That is, if one group is
- found to be superior  $(P \le .05)$ , the tipping point will identify the shift parameter necessary to
- yield P > .05. Conversely, if the null hypothesis is not rejected (P > .05), two tipping points will
- be identified one that would make aflibercept superior and one that would make bevacizumab
- + deferred aflibercept superior. In either case, this tipping point will be evaluated to determine if
- it is plausible. If not, then the MAR assumption is likely reasonable. For example, if the tipping
- 78 point were 100 letters, then this would be evidence that the MAR assumption is reasonable.

### Per-Protocol Analysis

- A per-protocol analysis will be conducted to estimate the treatment effect for each group among
- 81 those not receiving any alternative treatment for DME (e.g., intravitreal corticosteroids). This
- 82 analysis will include observed data from all randomized up to the time of alternative treatment
- 83 for DME. Data collected after the alternative treatment will be set to missing prior to imputation.
- 84 Imputation will otherwise be similar to the primary analysis. Note that focal/grid laser is allowed
- only if failure criteria have been met. The intention-to-treat analysis is considered the primary
- analysis. If the results of the primary and per-protocol analyses differ substantially, then
- 87 exploratory analyses will be performed to evaluate factors that may have contributed to the
- difference. The per-protocol analysis will only be performed if more than 10% of randomized
- 89 participants would be excluded by these criteria.

### Confounding Analysis

- Imbalances between groups in important covariates are not expected to be of sufficient
- magnitude to produce confounding in the primary analysis. However, the presence of
- 93 confounding in the primary analysis will be evaluated in additional regression models using
- observed data (no imputation) by including baseline participant and study eye covariates
- 95 including but not limited to the following:
- 96 Age

79

90

97

99

102

106

- Duration of diabetes
- 98 HbA1c
  - Mean arterial blood pressure
- 100 Prior PRP
- Prior treatment for DME
  - Diabetic retinopathy severity level on fundus photographs as graded by the reading center
- Each of the following within 500 μm of the center of the macula on OCT as graded by the reading center (minimum 20 eyes in the cohort with and without the characteristic):
- 105 o Epiretinal membrane
  - Vitreomacular traction
  - Cystoid abnormalities
- 108 o Subretinal fluid

- Each of the following within 1800 μm of the center of the macula on fundus photography as graded by the reading center (minimum 20 eyes in the cohort with and without the characteristic):
  - Hemorrhages/microaneurysms
- 113 o Hard exudates

114

120

- Surface wrinkling retinopathy
- Additional variables associated with the outcome will be included in regression models if there is
- an imbalance in the variables between treatment groups. Imbalance by treatment group will not
- be judged using statistical testing. Instead, imbalance will be judged by whether the size of the
- imbalance is clinically important, i.e., whether the imbalance is large enough to have a clinically
- important effect on the primary outcome.

### 2.2 Subgroup Analyses

- Pre-planned subgroup analyses will repeat the primary analysis while including an interaction
- term for the baseline subgroup factor by treatment. Missing data will be imputed by treatment
- group similarly to the primary analysis except that the subgroup factor will be included in the
- imputation model.<sup>1</sup>
- 125 A significant  $(P \le .05)$  type III test of the interaction term will be taken as an indication that
- subgroup effects need to be explored for full interpretation of the trial results. It is recognized
- that the study is not powered to detect subgroup effects and that lack of significance for the
- subgroup tests of interaction is not necessarily an indication that subgroup effects do not exist.
- 129 Interpretation of subgroup analyses will depend on whether the overall analysis demonstrates a
- significant treatment effect. In the absence of a significant treatment effect in the primary
- analysis, subgroup analyses will be interpreted with caution.
- Baseline variables to be evaluated for subgroup effects include the following:
- OCT central subfield thickness:  $< 400 \mu m \text{ vs} \ge 400 \mu m$  (Stratus equivalent)
- Visual acuity: 20/50 to 20/63 vs. 20/80 to 20/320
- Subgroups will only be analyzed if there are at least 20 eyes in each treatment group for each
- subgroup to increase statistical precision. Cutoffs of continuous outcomes may be modified to
- achieve a reasonable number of eyes in each group.
- The above subgroups are considered of primary interest. For each variable, the rationale for
- performing the analysis is listed in Table 1 below.

### Table 1. Subgroup analyses.

140

| Variable | Rationale |
|---|---|
| OCT central subfield thickness | Eyes with greater OCT central subfield thickness may have higher anti-<br>VEGF levels, leading to a larger relative treatment effect for the drug<br>with stronger VEGF binding affinity (aflibercept). |
| Baseline visual acuity | Eyes with lower visual acuity may have higher VEGF levels, leading to a larger relative treatment effect for the drug with stronger VEGF binding affinity (aflibercept). |

- 141 The following subgroup factors will be evaluated in exploratory analyses. Only point estimates
- and 95% confidence intervals for the within-subgroup treatment effects will be presented -P
- values will not be presented. The finding of a subgroup effect for any of these factors will be
- interpreted as hypothesis generating only and in need of confirmation from further studies.
- Prior treatment for DME: yes vs. no
- 146 HbA1c: < 7.5% vs.  $\ge 7.5\%$
- Sex: female vs. male
- Race/Ethnicity: Non-Hispanic White vs. Non-Hispanic Black/African American vs.
- Hispanic or Latino (exclude all other groups due to anticipated small sample size)

### 150 **2.3 Center Effects**

- 151 The number of study participants per center is expected to be small for many centers. Therefore,
- center effects will not be included in the statistical model. However, for centers with a large
- number of study participants ( $N \ge 20$  in either treatment group), heterogeneity across centers will
- be explored using random center effects by estimating empirical best linear unbiased predictors
- along with 95% confidence intervals.

### 3.0 Secondary Outcome Analyses

### 3.1 Visual Acuity and OCT

- Additional analyses of visual acuity will use the imputed data sets created for the primary
- outcome. For OCT outcomes, new imputed data sets will be created similarly by substituting
- baseline central subfield thickness (converted to a common scale based on the most accurate
- 161 conversion algorithms available) and change in central subfield thickness from baseline for
- baseline visual acuity and change in visual acuity from baseline, respectively. A plot of mean
- 163 change in OCT central subfield thickness over time by group will be constructed using observed
- 164 data.

156

- Analyses will be conducted at 24, 52 and 104 weeks unless otherwise noted. P values will be
- calculated for mean change in visual acuity and mean change in OCT central subfield thickness
- at 104 weeks only. All other secondary outcomes will be summarized with a model-based point
- estimate and 95% between-group confidence interval (no P value).

169 Analyses of continuous outcomes will be conducted in a manner similar to the primary analysis using linear mixed effects models and substituting central subfield thickness for visual acuity, 170 171 depending on the outcome.

Analyses of binary outcomes will be conducted using binomial regression with an identity link (estimating risk difference),<sup>2</sup> robust variance estimation, and adjustment for baseline visual acuity or OCT central subfield thickness (depending on the outcome). Generalized estimating equations (GEE) will be used to control for correlations arising from participants contributing two study eyes to the analysis. Baseline visual acuity (for visual acuity outcomes) or central subfield thickness (for central subfield thickness outcomes) and the number of study eyes will be included as covariates. The proportion of eyes meeting the outcome at the visit will be reported for each treatment group. In addition, the between-group risk difference and 95% confidence interval for the treatment effect will be presented; the P value will not be presented. If binomial regression fails to converge in one or more outcomes, then logistic regression with a random intercept for participant, conditional standardization, and the delta method (to estimate the risk difference)<sup>3</sup> may be used instead for all binary outcomes.

### Table 2. Analyses of Secondary Visual Acuity and OCT Outcomes.

172

173

174 175

176

177

178

179

180

181

182 183

184

188

189

| Outcome | Analysis Technique |
|---|---|
| Mean change in visual acuity from baseline | Linear mixed model <sup>a</sup> |
| Success proportion: visual acuity gain ≥ 15 letters | Binomial regression with GEE b |
| Success proportion: visual acuity gain ≥ 10 letters | Binomial regression with GEE <sup>b</sup> |
| Failure proportion: visual acuity loss ≥ 10 letters | Binomial regression with GEE <sup>b</sup> |
| Failure proportion: visual acuity loss ≥ 15 letters | Binomial regression with GEE b |
| Success proportion: visual acuity ≥ 84 letters (~20/20) | Binomial regression with GEE b |
| Success proportion: visual acuity ≥ 69 letters (~20/40) | Binomial regression with GEE b |
| Failure proportion: visual acuity ≤ 38 letters (~20/200) | Binomial regression with GEE b |
| Mean change in OCT central subfield thickness from baseline | Linear mixed model <sup>a</sup> |
| Proportion of eyes with OCT central subfield thickness below the gender-specific spectral domain OCT threshold for CI-DME <sup>c</sup> | Binomial regression with GEE <sup>b</sup> |
| Mean change in OCT retinal volume from baseline | Linear mixed model <sup>b</sup> |

<sup>185</sup> <sup>a</sup> At 24 and 52 weeks, a point estimate and 95% CI will be provided, but a P value will not be provided. At 104 186 weeks, a P value will be provided only if the primary analysis demonstrates a significant difference. 187

<sup>&</sup>lt;sup>b</sup> A point estimate and 95% CI will be provided, but a P value will not be provided.

<sup>&</sup>lt;sup>c</sup> For Zeiss Cirrus,  $\geq 290 \mu m$  for women and  $\geq 305 \mu m$  for men. For Heidelberg Spectralis,  $\geq 305 \mu m$  for women and ≥ 320 µm for men. No imputation for this outcome because the threshold values are machine specific and not Stratus equivalents, which are being imputed.

### 3.2 Changes in Diabetic Retinopathy

191

192

193194

195

196

197

198

199

200

201

203

204

206

207

The proportion of eyes with 2-step improvement or worsening of diabetic retinopathy on fundus photographs (defined in Table 3) will be assessed at 52 and 104 weeks using observed data only (no imputation). Analyses will be conducted with binomial regression while adjusting for baseline diabetic retinopathy severity (ordinal transformation) and using GEE to control for the correlation arising from participants contributing two study eyes to the analysis. Baseline ordinal diabetic retinopathy severity and the number of study eyes will be included as covariates. The proportion of eyes meeting the outcome at the visit will be reported for each treatment group. In addition, the risk difference and 95% confidence interval for the treatment effect will be reported, but not a *P* value.

Table 3. Definitions of Diabetic Retinopathy Improvement and Worsening for Eyes

| Baseline | | Worsening<br>(if follow up ≥) | Improvement<br>(if follow up ≤) |
|---|---|---|---|
| | 10/12 | 35 | Exclude |
| | 14/15/20 | 43 | Exclude |
| NPDR | 35 | 47 | 10/12 |
| NPDK | 43 | 53 | 14/15/20 |
| | 47 | 61 | 35 |
| | 53 | 61 | 43 |
| | 61 | 71 | 53 |
| | 65 | 75 | 53 |
| PDR | 71 | 81 | 61 |
| PDK | 75 | 81 | 65 |
| | 81 | Exclude | 71 |
| | 85 | Exclude | 75 |

Abbreviations: NPDR, non-proliferative diabetic retinopathy; PDR, proliferative diabetic retinopathy.

### 3.3 Additional Secondary Outcomes

Additional secondary outcomes will be evaluated 104 weeks, unless otherwise specified below.

### 205 Table 4. Additional Secondary Outcomes.

| Outcome | Analysis Technique <sup>a</sup> |
|---|---|
| Time to receipt of panretinal photocoagulation, vitrectomy, or occurrence of vitreous hemorrhage, traction retinal detachment, neovascularization of the iris, or neovascular glaucoma <sup>b</sup> | Marginal Cox proportional hazards regression |
| Number of injections up to the visit ° | Linear mixed model (52 and 104 weeks) |
| Number of visits <sup>d</sup> | Independent samples t-test |

<sup>&</sup>lt;sup>a</sup> Point estimates and 95% confidence intervals will be presented, but P values will not be presented.

<sup>&</sup>lt;sup>b</sup> Includes all randomized eyes, regardless of visit completion, and all visits up to and including the 104-week visit

- <sup>c</sup>Limited to eyes that complete the visit or any later common visit
- 209 d Evaluated at 104 weeks for 104-week completers among participants with one study eye. Bilateral participants are
- 210 excluded because number of visits is a participant-level outcome and treatment group is an eye-level variable.
- 211 Kaplan-Meier estimates for the time to receipt of panretinal photocoagulation, vitrectomy or
- occurrence of vitreous hemorrhage, traction retinal detachment, neovascularization of the iris, or
- 213 neovascular glaucoma will be provided. A marginal Cox proportional hazards model with a
- 214 robust sandwich estimate of the covariance matrix will be used to control for correlations arising
- 215 from bilateral participants. Baseline ordinal diabetic retinopathy severity and the number of
- 216 study eyes will be included as covariates. The model will adjust for ordinal baseline diabetic
- 217 retinopathy severity because these events all represent worsening of diabetic retinopathy, and
- eyes with more advanced diabetic retinopathy at baseline are more likely to experience
- worsening. The treatment effect will be measured as a hazard ratio and will be reported with the
- associated 95% confidence interval, but not a P value. When the number of events is low (i.e.,
- less than 10 in either treatment group), these time-to-event analyses will be replaced by
- comparing the percentage in each treatment group with the PDR event at any time during follow-
- 223 up. A 95% confidence interval on the difference in proportions will be calculated by inverting
- 224 two separate one-sided exact tests that are based on the score statistic.
- For comparison of the number of injections, a linear mixed model will be used with the number
- of study eyes included as a covariate. For comparison of the number of visits, an independent
- samples t-test limited to participants with one study eye will be used.

### **4.0 Outcomes within Treatment Groups**

- Within each treatment group, the following outcomes will be tabulated without formal statistical comparisons.
  - Distribution and mean (standard deviation) number of intravitreous injections performed up to 24, 52, and 104 weeks as well as the intervening periods for eyes completing any common visit at or beyond the upper limit (e.g., for injections through 52 weeks, eyes must have completed the 52-, 68-, 84-, or 104-week visit).
    - o Intervals will be closed on the left and open on the right (e.g., for injections through 24 weeks, an injection given at 24 weeks will not be counted towards the total; however, an injection given at 24 weeks will count for the interval of 24 to 52 weeks), unless the upper boundary is at 104 weeks in which case the interval is closed on the left and right.
    - Proportion of eyes that met switch criteria by the 12, 24, 52, or 104-week visits.
      - Estimated using the Kaplan-Meier method.

### **5.0 Economic Analysis**

231

232

233234

235

236237

238

239

240

- The purpose of the economic analysis is to compare the treatment groups with respect to cost. An
- incremental cost effectiveness ratio (ICER) will be calculated. Data from the clinical trial on the

245 number of clinic visits completed, number of procedures performed (e.g., OCT, fundus 246 photographs), and number of aflibercept and bevacizumab treatments will be used to estimate an 247 average cost per patient for each treatment arm. The Medicare Fee Schedule will be used to 248 estimate medical costs. For outcomes measured at the participant level, bilateral participants are 249 non-informative with respect to the treatment comparison and will not be included in the 250 economic analyses. 251 **6.0 Safety Analysis** 252 Adverse events will be categorized as study eye, fellow eye, or systemic. A full listing of adverse 253 events will be tabulated by treatment. An additional tabulation will be made for adverse events 254 possibly related to study treatment. 255 All randomized eyes will be included in the safety analysis and analyzed according to treatment 256 assignment at randomization, regardless of treatment actually received. Any adverse event that 257 occurred up to and including the 104-week visit (or, if the participant did not complete the 104-258 week visit, 896 days from randomization, the end of the 2-year analysis window) will be 259 reported. 260 **6.1 Study Eye Adverse Events** 261 The frequency of the event occurring at least once will be calculated for study eyes in each 262 treatment group. The proportion of eyes experiencing each outcome will be compared between 263 treatment groups using Barnard's unconditional exact test, considering the number of eyes in 264 each treatment group fixed. It is noted that this method does not adjust for the potential correlation arising from participants with two study eyes; however, given the low expected 265 266 frequency of adverse events and small proportion of bilateral subjects, the impact should be 267 minimal. Adjustment for such correlations would be statistically problematic due to the low 268 frequency of events. 269 The following ocular adverse events will be assessed: 270 o Endophthalmitis 271 o Retinal detachment (rhegmatogenous, traction, combined rhegmatogenous and traction, or not otherwise specified) 272 273 Rhegmatogenous retinal detachment (tabulated without formal analysis) 274 Traction retinal detachment (tabulated without formal analysis) 275 o Traumatic cataract due to intravitreous injection 276 Analysis limited to eyes with phakic lens at baseline 277 Vitreous hemorrhage

o Ocular inflammation

279 o Intraocular pressure (IOP) elevation (composite outcome; individual components below will be tabulated without formal analysis): 280 281 Increase in IOP  $\geq$  10 mmHg from baseline (at a follow-up visit) 282  $IOP \ge 30 \text{ mmHg}$  (at a follow-up visit) Initiation of medication to lower IOP that was not in use at baseline 283 284 Glaucoma procedure 285 Neovascularization of the iris 286 o Neovascular glaucoma 287 **6.2 Systemic Adverse Events** 288 Systemic adverse events will be reported in three groups: (1) unilateral participants randomized 289 to bevacizumab + deferred aflibercept, (2) unilateral participants randomized to aflibercept, and (3) bilateral participants randomized to bevacizumab + deferred aflibercept in one eye and 290 291 aflibercept in the other eye. The frequency of each event occurring at least once per participant will be calculated. The proportion of participants with each systemic adverse event will be 292 293 compared among groups using Fisher's exact test. If the overall test has  $P \le 0.05$ , then pairwise 294 comparisons between groups will be conducted using Fisher's exact test without the need to adjust for multiple comparisons.<sup>5</sup> The following systemic adverse events will be assessed: 295 296 o Primary: 297 Death 298 Serious adverse event 299 Hospitalization 300 Cardiovascular and cerebrovascular events according to the Antiplatelet 301 Trialists' Collaboration (excerpted from BMJ Jan 8, 1994): 302 • Nonfatal myocardial infarction 303 Nonfatal stroke (counted only if symptoms lasted at least 24 hours) 304 • Death attributed to cardiac, cerebral, hemorrhagic, embolic, other vascular (does not need to be ischemic in origin), or unknown cause 305 306 • At least one event (nonfatal myocardial infarction, nonfatal stroke, or 307 death attributed to potential vascular or unknown cause) 308 Note that transient ischemic attack, angina, possible myocardial infarction, and possible stroke 309 are not counted. Nonfatal myocardial infarction and nonfatal stroke require that the patient be 310 alive at the end of the study. If not, then only the death is counted.

| 311 | <ul> <li>Secondary (for tabulation without statistical comparison):</li> </ul> |
|---|---|
| 312<br>313 | <ul> <li>Frequency of at least one event per participant in each Medical Dictionary for<br/>Regulatory Activities (MedDRA) system organ class</li> </ul> |
| 314 | 7.0 Additional Tabulations |
| 315 | The following will be tabulated according to treatment group: |
| 316 | Baseline demographic and clinical characteristics |
| 317 | • Visit completion rate for each annual visit (excluding deaths) |
| 318 | Treatment adherence |
| 319 | 8.0 General Principles for Analysis |
| 320 | 8.1 Analysis Cohort |
| 321<br>322<br>323 | Unless otherwise stated, all treatment comparison analyses will follow the intention-to-treat principle with all randomized eyes included and each eye analyzed according to the randomized treatment assignment, regardless of treatment actually received. |
| 324 | 8.2 Visit Windows for Analysis |
| 325<br>326<br>327<br>328 | For common visits, the analysis windows will be defined according to Table 5. Note that all eyes have visits every 4 weeks in year 1, but the protocol visit schedule varies in year 2 depending on the clinical course. Therefore, visit windows at 68 and 84 weeks have been defined for analysis purposes. |
| 329<br>330 | If multiple visits fall within the same analysis window, the following algorithm will be used to prioritize which visit will be used for analysis: |
| 331 | • Visits with non-missing visual acuity data will be prioritized over visits with missing data |
| 332<br>333 | • If there is no protocol visit in the analysis window, then the visit closest to the target will be used |
| 334<br>335 | o For visits falling in more than one window, priority will be given to the 24-, 52-, and 104-week visits. Otherwise, the visit will be assigned to the earlier window |

**Table 5. Analysis Windows for Outcome Visits** 

| Protocol Visit | Target | Analysis Window | |
|----------------|----------|-----------------|----------------------------|
| 4 weeks | 28 days | 14 – 42 days | $(4 \pm 2 \text{ weeks})$ |
| 8 weeks | 56 days | 42 – 70 days | $(8 \pm 2 \text{ weeks})$ |
| 12 weeks | 84 days | 70 – 98 days | $(12 \pm 2 \text{ weeks})$ |
| 16 weeks | 112 days | 98 – 126 days | $(16 \pm 2 \text{ weeks})$ |
| 20 weeks | 140 days | 126 – 154 days | $(20 \pm 2 \text{ weeks})$ |
| 24 weeks | 168 days | 154 – 182 days | $(24 \pm 2 \text{ weeks})$ |
| 28 weeks | 196 days | 182 – 210 days | $(28 \pm 2 \text{ weeks})$ |
| 32 weeks | 224 days | 210 – 238 days | $(32 \pm 2 \text{ weeks})$ |
| 36 weeks | 252 days | 238 – 266 days | $(36 \pm 2 \text{ weeks})$ |
| 40 weeks | 280 days | 266 – 294 days | $(40 \pm 2 \text{ weeks})$ |
| 44 weeks | 308 days | 294 – 322 days | $(44 \pm 2 \text{ weeks})$ |
| 48 weeks | 336 days | 322 – 350 days | $(48 \pm 2 \text{ weeks})$ |
| 52 weeks | 364 days | 308 – 420 days | $(52 \pm 8 \text{ weeks})$ |
| 68 weeks | 476 days | 420 – 532 days | $(68 \pm 8 \text{ weeks})$ |
| 84 weeks | 588 days | 532 – 644 days | (84 ± 8 weeks) |
| 104 weeks | 728 days | 644 – 896 days | (92–128 weeks) |

### 8.3 Missing Data

In general, the strategy for handling missing data is included with the description of each individual analysis. Where not otherwise specified, only participants with non-missing data are included in the analysis.

### 8.4 Outliers

To help ensure that statistical outliers do not have undue impact on analyses of continuous visual acuity and OCT outcomes (including the primary outcome), change in visual acuity change in central subfield thickness, and change in retinal volume will be truncated to  $\pm$  3 standard deviations. The standard deviations will be based on observed data from 104-week completers at the 104-week visit, irrespective of treatment group. Truncation will be performed after imputation of missing data, where applicable (i.e., raw data will be used for imputation). For the primary outcome, AUC will be calculated based on the imputed values after truncation. There will be no truncation of the AUC outcome itself.

### 8.5 Model Assumptions

All model assumptions, including linearity, normality of residuals, heteroscedasticity, and proportional hazards will be verified. If model assumptions are not reasonably satisfied, then covariates may be categorized or excluded, and a nonparametric approach, transformation, or robust method may be considered.

```
8.6 Multiple Testing
356
      The primary analysis will be conducted at alpha of 0.05. If the primary analysis demonstrates a
357
      significant treatment group difference, then mean change in visual acuity from baseline at 104
      weeks and mean change in OCT central subfield thickness from baseline at 104 weeks will be
358
359
      tested as secondary outcomes. The Holm method will be used to provide strong control of alpha
360
      at 0.05.5 If the primary analysis fails to show a significant difference, then outcomes will be
361
      described with summary statistics, model-based point estimates, and between-group 95%
362
      confidence intervals without a P value. This approach controls the family-wise error rate at 5%.
363
      There will be no formal adjustment for multiplicity in sensitivity, subgroup, or safety analyses.
      For exploratory subgroup analyses, the number of significant results expected by chance given
364
365
      the number of comparisons will be noted.
366
      9.0 Example SAS Code
367
      Below is an example of SAS code for the primary outcome analysis. The actual code used might
368
      differ due to variable naming conventions.
369
      /* Generate Imputed Data Sets */
370
      proc mi data=studyEyes nimpute=100 seed=9999 out=outMI;
371
         var va0 vaChg4 vaChg8 vaChg12 vaChg16 vaChg20 vaChg24 vaChg28
372
             vaChg32 vaChg36 vaChg40 vaChg44 vaChg48 vaChg52 vaChg68
373
             vaChg84 vaChg104 switchGrpFlg bilateralFlg;
374
      run;
375
      /* ...DATA steps to truncate changes in visual acuity and calculate primary
376
      outcome (vaChgAUC104)... */
377
      /* Linear Mixed Model for Each Imputation */
378
      proc mixed data=outMI empirical;
379
         by imputation;
380
         class PtID;
381
         model vaChgAUC104=va0 bilateralFlg switchGrpFlg / solution
382
           covb ddfm=kr2;
383
         random int / subject=PtID;
384
         ods output solutionF=mixParms covb=mixCovB;
385
      run;
```

```
/* Combine Results */
proc mianalyze data=mixParms covb(effectvar=rowcol)=mixCovB

edf=308;

/* 312 eyes minus 3 fixed effects + intercept = 308 degrees of freedom */
modeleffects va0 bilateralFlg switchGrpFlg;

run;
```

### **392 10.0 References**

- 393 1. Sullivan TR, White IR, Salter AB, Ryan P, Lee KJ. Should multiple imputation be the method of choice for handling missing data in randomized trials? *Stat Methods Med Res.* 395 2018;27(9):2610-2626.
- 396 2. Spiegelman D, Hertzmark E. Easy SAS calculations for risk or prevalence ratios and differences. *Am J Epidemiol.* 2005;162(3):199-200.
- 398 3. Localio AR, Margolis DJ, Berlin JA. Relative risks and confidence intervals were easily computed indirectly from multivariable logistic regression. *J Clin Epidemiol*. 2007;60(9):874-882.
- 401 4. Lee EW, Wei LJ, Amato DA. Cox-type regression analysis for large numbers of small groups of correlated failure time observations. Dordrecht: Kluwer Academic; 1992.
- Dmitrienko A, D'Agostino RB, Sr. Multiplicity Considerations in Clinical Trials. N Engl
   J Med. 2018;378(22):2115-2122.